CLINICAL TRIAL: NCT00219856
Title: Prospective, Randomized, Simple Blind Study Comparing the Effects of an Anaesthesia With Propofol to an Anaesthesia With Desflurane on Oxydative Stress and Liver Function Recovery After Hepatectomy
Brief Title: Effects of Propofol on Oxidative Stress and Liver Regeneration After Partial Hepatectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Direction of Clinical Research, Rennes University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFSSAPS 040366; PHRC/03-02 (Other: Rennes University Hospital); CIC0203/026
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Hepatectomy
Keywords: Propofol; Hepatectomy; Oxidative stress
MeSH Terms: interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Anesthesic induction and maintenance with intravenous propofol.
  Interventions: Drug: Propofol
- 2 (Active Comparator): Anesthesic induction with intravenous penthotal and maintenance with inhaled desflurane.
  Interventions: Drug: Penthotal; Drug: Desflurane

INTERVENTIONS:
Drug: Propofol — * Induction : intravenous propofol aiming a concentration of 4 to 8 µg/ml
  * Maintenance : intravenous propofol aiming a concentration of 3 to 6 µg/ml
  Arms: 1
Drug: Penthotal — Intravenous penthotal at the dose of 3 to 5 mg/kg
  Arms: 2
Drug: Desflurane — Inhaled desflurane aiming an alveolar concentration of 4 to 6 per cent.
  Arms: 2

SUMMARY:
Propofol is an anaesthetic agent that showed in vitro and in vivo anti oxidant properties. No data are available concerning the potential benefit of a total anaesthesia with propofol in partial hepatic surgery. Patients who undergo partial hepatic resection have frequent liver insufficiency that could be related in part to the oxidative stress induced by clamping the hepatic vessels during the surgical intervention. Our hypothesis is that propofol, by increasing liver resistance to this ischemia-reperfusion phenomenon, could improve the remaining liver function recovery, and therefore could reduce post surgical morbidity.

The aim of the study is to evaluate the anti oxidant effects of propofol compared to another widely used anaesthetic agent, inhaled desflurane, during and after partial hepatic resection with hepatic vessels clamping. The primary endpoint will be the level of malondialdehyde (a plasmatic marker of oxidative stress), 30 minutes after the end of hepatic clamping.

DETAILED DESCRIPTION:
Propofol is an anaesthetic agent that showed in vitro and in vivo anti oxidant properties. No data are available concerning the potential benefit of a total anaesthesia with propofol in partial hepatic surgery. Patients who undergo partial hepatic resection have frequent liver insufficiency that could be related in part to the oxidative stress induced by clamping the hepatic hilum during the surgical intervention. Our hypothesis is that propofol, by increasing liver resistance to ischemic-reperfusion injury, could improve the remaining liver function recovery, and therefore could reduce post surgical morbidity.

The aim of the study is to evaluate the anti oxidant effects of propofol compared to another widely used anaesthetic agent, inhaled desflurane, during and after partial hepatic resection with hepatic hilum clamping.

The primary endpoint will be the level of malondialdehyde (a plasmatic marker of oxidative stress), 30 minutes after the end of hepatic clamping.

The evolution over time of other markers of oxidative stress will be studied (glutathione, myeloperoxidase, nitric oxide), as well as functional and biological markers of liver regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* Need for partial hepatic resection requiring heptic clamping
* Resection of 4 liver segments or less
* In case of cirrhosis, child A
* Written informed consent

Non-inclusion Criteria:

* Hemochromatosis
* chemotherapy in the previous week before inclusion
* Thrombosis of the portal vein or the hepatic artery
* Absence of contraception among fertil woman
* Concomitant treatment that could have potential interaction with propofol
* Concomitant treatment known to have antioxidant properties
* Inclusion in another study protocol using a medication incompatible with the present study
* Patient in which the follow up seems impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-08; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Plasma MDA levels | 30 minutes after the end of hepatic clamping

SECONDARY OUTCOMES:
Kinetics of post surgical biological hepatic function recovery | Days 1, 2, 5, 10
  * Gamma gluatamyltransferase
  * ASAT
  * ALAT
  * Factor V
  * AlfagluthationeS-transferase
Kinetics of post surgical hepatic function recovery | Day 2
  Monoethylglycinexylidide (MEGX) test
Other biological markers of oxidative stress | Days 1 and 2
  * Glutathione
  * Myeloperoxidase
  * Nitric oxide
Hemodynamics during and after surgery | Days 1 and 2
  * Mean arterial pressure
  * Heart rate
  * Diuresis
Surgery related complications | 10 days
  * Liver insufficiency
  * Hepato renal syndrome
  * Local infections

CONTACTS AND LOCATIONS:
Overall Officials: David Aguillon, MD, Principal Investigator — Rennes University Hospital; Yannick Malledant, MD, Study Director — Rennes University Hospital; Bruno Laviolle, MD, Study Chair — Rennes University Hospital
Locations (1):
- Surgical Intensive Care Unit - Rennes University Hospital, Rennes, France